CLINICAL TRIAL: NCT01831089
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination With Weekly Paclitaxel, With or Without Bevacizumab, in Patients With Selected Advanced Solid Tumors
Brief Title: Phase I Study of Lurbinectedin (PM01183) in Combination With Paclitaxel, With or Without Bevacizumab, in Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-007-13
Record Dates: First submitted 2013-04-02; First posted 2013-04-15 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Ovarian Cancer; Gynecological Cancer; Head and Neck Carcinoma; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Non-squamous Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): PM01183 + paclitaxel +/- bevacizumab
  Interventions: Drug: PM01183 + paclitaxel +/- bevacizumab

INTERVENTIONS:
Drug: PM01183 + paclitaxel +/- bevacizumab — PM01183: 1 mg and 4 mg vials. Powder for concentrate for solution for infusion
  paclitaxel: 6 mg/ml concentrate for solution for infusion
  bevacizumab: 25 mg/ml concentrate for solution for infusion
  Once a recommended dose is defined for the PM01183 and weekly paclitaxel combination, the feasibility of adding bevacizumab to this combination will be explored in a prospectively selected cohort of patients

SUMMARY:
Clinical trial of PM01183 in combination with paclitaxel, with or without bevacizumab, in patients with solid tumors

DETAILED DESCRIPTION:
Clinical trial to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM01183 in combination with weekly paclitaxel, with or without bevacizumab. Once a recommended dose is defined for the PM01183 and weekly paclitaxel combination, the feasibility of adding bevacizumab to this combination will be explored in a selected cohort of patients to characterize the safety profile and feasibility of this combination, to obtain preliminary information on antitumor activity, to obtain preliminary information on quality of life (QoL), to characterize the pharmacokinetics (PK) of this combination and to detect major drug-drug PK interactions and PK(pharmacokinetic)/PD(pharmacodynamic) correlation and to conduct an exploratory pharmacogenomic(PGx) analysis in patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated written informed consent
* Age between 18 and 75 years old (both inclusive)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 1
* Life expectancy ≥ 3 months.
* Patients with a histologically/cytologically confirmed diagnosis of advanced and/or unresectable disease of any of the following tumors:

  1. Breast cancer
  2. Epithelial ovarian cancer or gynecological cancer
  3. Head and neck squamous cell carcinoma
  4. Non-small cell lung cancer
  5. Small cell lung cancer
  6. Platinum-refractory germ-cell tumors.
  7. Adenocarcinoma or carcinoma of unknown primary site
* Adequate bone marrow, renal, hepatic, and metabolic function
* Recovery to grade ≤ 1 or to baseline from any Adverse Event (AE) derived from previous treatment (excluding alopecia of any grade).
* Pre-menopausal women must have a negative pregnancy test before study entry and agree to use a medically acceptable method of contraception throughout the treatment period and for at least six weeks after treatment discontinuation

Exclusion Criteria:

* Prior treatment with PM01183 or weekly paclitaxel or nanoalbumin-paclitaxel
* Patients who have previously discontinued paclitaxel-based regimes due to drug related toxicity.
* Known hypersensitivity to bevacizumab or any component of its formulation
* Patients who have previously discontinued bevacizumab-containing regimes due to drug-related toxicity.
* More than three prior lines of chemotherapy
* Less than three months since last taxane-containing therapy.
* Wash-out period:

  1. Less than three weeks since the last chemotherapy-containing regimen
  2. Less than three weeks since the last radiotherapy dose
  3. Less than four weeks since last monoclonal antibody-containing therapy
* Concomitant diseases/conditions:

Unstable angina, myocardial infarction, valvular heart disease, encephalopathy, ischemic attacks, hemorrhagic or ischemic cerebrovascular accident (CVA) or ongoing pulmonary embolism within last year, arrhythmia, hepatopathy, uncontrolled infection, hemoptysis or oxygen requiring dyspnea, known HIV infection, bleeding risk, muscular problems, peripheral neuropathy, Symptomatic or progressive brain metastases or leptomeningeal disease.

* Men or pre-menopausal women who are not using an effective method of contraception as previously described; actively breast feeding women.
* Patients who have pelvic irradiation with doses ≥ 45 Grays (Gy).
* History of previous bone marrow and/or stem cell transplantation.
* Confirmed bone marrow involvement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- New York, New York, United States
- Madrid, Spain
- Bellinzona, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 69 patients were enrolled at 3 investigational sites: 55 Group A (paclitaxel plus PM01183) and 14 Group B (paclitaxel+PM01183 and BEV). Patients participated in this trial between 15/Oct/2013 and 14/Jul/2016 (last FU). The first dose of the first cycle was given on 23/Oct/2013 and the last dose of the last cycle was given on 23/Jun/2016
Pre-assignment Details: Signed IC,Age 18-75,ECOG PS≤1,Life expectancy≥3 months,Histologically/cytologically confirmed diagnosis of advanced and/or unresectable disease according to the groups,adequate status patient,no AEs,negative pregnancy test.
Groups:
- Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD]: Cohort I
  * Paclitaxel 60.0 mg/m2 as an i.v. infusion on Days 1, 8 and 15 q3wk, over one hour via a central or peripheral venous catheter through a pump device with an appropriate infusion line and filter.
  * PM01183 3.0 mg FD as an i.v. infusion on Day 1 q3wk, after paclitaxel infusion, over one hour via a central catheter (or over a minimum dilution of 250 mL if a peripheral venous catheter was used) through a pump device.
  Patients in this group were to receive paclitaxel and PM01183 for up to six cycles, in the absence of disease progression or unacceptable toxicity; then, PM01183 could be continued alone until progression, unacceptable toxicity, patient's decision, or Investigator's decision upon the Sponsors' agreement.
- Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD]: Cohort II
  * Paclitaxel 60.0 mg/m2 as an i.v. infusion on Days 1, 8 and 15 q3wk, over one hour via a central or peripheral venous catheter through a pump device with an appropriate infusion line and filter.
  * PM01183 4.0 mg FD as an i.v. infusion on Day 1 q3wk, after paclitaxel infusion, over one hour via a central catheter (or over a minimum dilution of 250 mL if a peripheral venous catheter was used) through a pump device.
  Patients in this group were to receive paclitaxel and PM01183 for up to six cycles, in the absence of disease progression or unacceptable toxicity; then, PM01183 could be continued alone until progression, unacceptable toxicity, patient's decision, or Investigator's decision upon the Sponsors' agreement.
- Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD: Cohort III
  * Paclitaxel 60.0 mg/m2 as an i.v. infusion on Days 1, 8 and 15 q3wk, over one hour via a central or peripheral venous catheter through a pump device with an appropriate infusion line and filter.
  * PM01183 5.0 mg FD as an i.v. infusion on Day 1 q3wk, after paclitaxel infusion, over one hour via a central catheter (or over a minimum dilution of 250 mL if a peripheral venous catheter was used) through a pump device.
  Patients in this group were to receive paclitaxel and PM01183 for up to six cycles, in the absence of disease progression or unacceptable toxicity; then, PM01183 could be continued alone until progression, unacceptable toxicity, patient's decision, or Investigator's decision upon the Sponsors' agreement.
- Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD]: Cohort IV
  * Paclitaxel 80.0 mg/m2 as an i.v. infusion on Days 1, 8 and 15 q3wk, over one hour via a central or peripheral venous catheter through a pump device with an appropriate infusion line and filter.
  * PM01183 5.0 mg FD as an i.v. infusion on Day 1 q3wk, after paclitaxel infusion, over one hour via a central catheter (or over a minimum dilution of 250 mL if a peripheral venous catheter was used) through a pump device.
  Patients in this group were to receive paclitaxel and PM01183 for up to six cycles, in the absence of disease progression or unacceptable toxicity; then, PM01183 could be continued alone until progression, unacceptable toxicity, patient's decision, or Investigator's decision upon the Sponsors' agreement.
- Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD]: Cohort V
  * Paclitaxel 80.0 mg/m2 as an i.v. infusion on Days 1, 8 and 15 q3wk, over one hour via a central or peripheral venous catheter through a pump device with an appropriate infusion line and filter.
  * PM01183 4.0 mg FD as an i.v. infusion on Day 1 q3wk, after paclitaxel infusion, over one hour via a central catheter (or over a minimum dilution of 250 mL if a peripheral venous catheter was used) through a pump device.
  Patients in this group were to receive paclitaxel and PM01183 for up to six cycles, in the absence of disease progression or unacceptable toxicity; then, PM01183 could be continued alone until progression, unacceptable toxicity, patient's decision, or Investigator's decision upon the Sponsors' agreement.
- Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg: All three study medications were administered via a central or a peripheral venous catheter through a pump device, as follows:
  * Paclitaxel 80.0 mg/m2 as an i.v. infusion on Days 1, 8 and 15 q3wk, over one hour.
  * PM01183 as an i.v. infusion on Day 1 q3wk, after paclitaxel infusion, over one hour.
  * Bevacizumab (BEV) 15 mg/kg as an i.v. infusion on Day 1 q3wk, immediately after paclitaxel and PM01183 infusions, Minimum duration of infusion was 90 minutes for the first dose and, if well tolerated, 60 minutes for the second dose and 30 minutes for all subsequent doses. nous catheter was used) through a pump device.
  Patients in this group were to receive paclitaxel, PM01183 and BEV for up to six cycles, in the absence of disease progression or unacceptable toxicity; then, both PM01183 and BEV could be continued until progression, unacceptable toxicity, patient's decision, or Investigator's decision upon the Sponsors' agreement.
Period: Cohort I: Dose Level 1
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 0 | 0 | 0 | 0 | 0
Period: Cohort II: Dose Level 2
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Started | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Clinical progressive disease | 0 | 1 | 0 | 0 | 0 | 0
Period: Cohort III: Dose Level 3
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Started | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 6 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Global end of study | 0 | 0 | 1 | 0 | 0 | 0
Period: Cohort IV: Dose Level 4
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Started | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 6 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 6 | 0 | 0
Period: Cohort V: Dose Level 5
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Started | 0 | 0 | 0 | 0 | 37 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 37 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 30 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Global end of study | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Period: Cohort B: Arm B
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 14
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Never treated | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Global end of study | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 37 | 14 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 6 | 5 | 23 | 12 | 51
  >=65 years | 1 | 0 | 0 | 1 | 14 | 2 | 18
Age, Continuous [Median (Full Range); unit: years] | 57 [53 to 72] | 50 [31 to 55] | 53.5 [41 to 63] | 46.5 [38 to 68] | 61.0 [38 to 74] | 57 [47 to 72] | 57 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 5 | 26 | 8 | 48
  Male | 1 | 0 | 2 | 1 | 11 | 6 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 1 | 2 | 1 | 1 | 6 | 1 | 12
  Spain | 2 | 1 | 3 | 4 | 12 | 6 | 28
  United States | 0 | 0 | 2 | 1 | 19 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD will be the lowest level at which one third or more evaluable patients experience a DLT in Cycle 1.
  DLTs are defined as AEs or laboratory abnormalities related to the study drugs occurred during Cycle 1.
Time Frame: The MTD was followed mainly during Cycle 1 through study completion, an average of 5 cycles for PM1183 in cohort A and 9.5 cycles in cohort B were observed (cycle duration: 3 weeks)
Population: Three patients at the RD were not evaluable because they did not receive a complete Cycle 1 due to disease-related grade 3 vomiting and early PD, disease-related grade 3 confusional state, and because not enough information for DLT evaluation was collected during Cycle 1.
Measure: Number; unit: mg/m2 / mg FD
Groups:
- Group A (Paclitaxel/PM01183): All participants who received at least 1 dose of Paclitaxel/PM01183, either at 60/3.0, 60/4.0, 60/5.0, 80/5.0, 80/4.0 mg/m2 / mg FD.
Arm/Group | Group A (Paclitaxel/PM01183)
Number analyzed (Participants) | 52
mg/m2 / mg FD | NA — Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD]

2. Primary Outcome: Recommended Dose (RD)
Description: The RD will be the highest DL explored with less than one third of the patients experiencing a DLT during Cycle 1.
  DLTs are defined as AEs or laboratory abnormalities related to the study drugs occurred during Cycle 1.
Time Frame: The RD was followed mainly during Cycle 1 through study completion, an average of 5 cycles for PM1183 in cohort A and 9.5 cycles in cohort B were observed (cycle duration: 3 weeks)
Population: as for outcome 1
Measure: Number; unit: mg/m2 / mg FD
Arm/Group | Group A (Paclitaxel/PM01183)
Number analyzed (Participants) | 52
mg/m2 / mg FD | NA — Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD]

3. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLTs are defined as AEs or laboratory abnormalities related to the study drugs occurred during Cycle 1.
Time Frame: DLT was followed mainly during Cycle 1 through study completion, an average of 5 cycles for PM1183 in cohort A and 9.5 cycles in cohort B were observed (cycle duration: 3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 34 | 12
Participants | 0 | 0 | 2 | 3 | 6 | 3

4. Secondary Outcome: Best Tumor Response
Description: Best overall response:Best response recorded from the start of the study treatment until the end of treatment Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to<10 mm Partial Response (PR):At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression) Stable Disease (SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum diameters while on study Treatment failure (TF):symptomatic deterioration or death due to progression
Time Frame: Through study completion, an average of 5 cycles for PM1183 in cohort A and 9.5 cycles in cohort B were observed (1 cycle =3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 33 | 10
Participants
  CR | 0 | 0 | 0 | 0 | 1 | 1
  PR | 1 | 0 | 2 | 4 | 12 | 4
  SD ≥3 months | 1 | 2 | 1 | 1 | 6 | 4
  SD <3 months | 0 | 0 | 1 | 0 | 1 | 0
  PD | 1 | 1 | 2 | 1 | 12 | 0
  Early PD | 0 | 0 | 0 | 0 | 1 | 0
  TF | 0 | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the date of first infusion of study treatment to the date of progression or death (due to any cause). If progression or death had not occurred at the time of the analysis, the PFS was censored.
Time Frame: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 33 | 10
months | 3.5 [1.7 to 5.6] | 3.1 [1.9 to 7.4] | 3.1 [1.0 to NA] — Not reached | 5.4 [1.7 to 8.8] | 3.9 [1.9 to 6.0] | 6.7 [2.4 to 9.3]

6. Secondary Outcome: Duration of Response (DR)
Description: Duration of response (DR) was defined as the time from the date when the response criteria (PR or CR, whichever was reached first) were fulfilled, to the first date when PD, recurrence or death was documented
Time Frame: as for outcome 4
Population: In cohort II, no patients with PR or CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Number analyzed (Participants) | 1 | 0 | 2 | 4 | 13 | 5
months | 1.6 [NA to NA] — Not reached |  | NA [2.0 to NA] — Not reached | 2.2 [0.9 to 4.7] | 4.1 [2.1 to 8.3] | 4.6 [1.4 to NA] — Not reached

7. Secondary Outcome: Quality of Life (QoL)
Description: Change from baseline to last cycle. European Organization for Research and Treatment of Cancer (EORTC) QLQ-C15-PAL scale scores.
  The EORTC QLQ-C15-PAL is an abbreviated 15-item version of the EORTC QLQ-C30 (version 3.0) developed for palliative care. Wilcoxon signed ranks test repeat-measure analyses of variance were used to measure the change value from baseline value. Data has to be analysed following the corresponding EORTC manual http://www.eortc.be/qol/files/SCManualQLQ-C15-PAL.pdf and the overall quality of life assessment is contained in 0 to 100 where a higher value represents a better state.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 26 | 8
score on a scale
  Pain | 5.6 (9.6) | 8.3 (11.8) | -13.3 (21.7) | 13.3 (13.9) | -4.2 (21.0) | 12.5 (30.5)
  Dyspnea | 0.0 (0.0) | 0.0 (47.1) | -6.7 (27.9) | 6.7 (14.9) | 11.1 (25.4) | 12.5 (24.8)
  Insomnia | 0.0 (33.3) | 16.7 (23.6) | 0.0 (0.0) | -6.7 (14.9) | 4.2 (34.5) | -12.5 (30.5)
  Appetite loss | -22.2 (38.5) | 0.0 (0.0) | -6.7 (14.9) | 0.0 (0.0) | 1.4 (30.3) | 16.7 (25.2)
  Constipation | 11.1 (19.2) | 0.0 (0.0) | 6.7 (14.9) | 13.3 (29.8) | -2.8 (23.9) | 8.3 (23.6)
  Overall QoL | 5.6 (9.6) | -16.7 (0.0) | -8.3 (21.5) | -6.7 (19.0) | -6.3 (22.4) | -10.4 (17.7)
  Physical functioning | -11.1 (19.2) | -6.7 (9.4) | -2.7 (6.0) | -13.3 (8.2) | -2.8 (19.8) | -8.3 (17.0)
  Fatigue | 3.7 (33.9) | 0.0 (0.0) | -2.2 (24.1) | 11.1 (13.6) | 6.5 (23.4) | 2.8 (22.0)
  Nausea / vomiting | -5.6 (9.6) | 8.3 (11.8) | 0.0 (11.8) | 3.3 (7.5) | 3.5 (9.8) | 2.4 (6.3)
  Emotional functioning | 16.7 (28.9) | -8.3 (35.4) | 0.0 (11.8) | 5.0 (33.1) | 6.3 (18.4) | 5.2 (16.0)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 cycles for PM1183 in cohort A and 9.5 cycles in cohort B were observed (1 cycle =3 weeks)
Description: In Group B: 14 patients were included, although only 12 were treated.
Arm/Group | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 3/37 | 2/14
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 3/6 | 2/6 | 15/37 | 7/14
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 6/6 | 36/37 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] (N=3) | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] (N=3) | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD (N=6) | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] (N=6) | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] (N=37) | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg (N=14)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel [60.0 mg/m2] / PM01183 [3.0 mg FD] (N=3) | Paclitaxel [60.0 mg/m2] / PM01183 [4.0 mg FD] (N=3) | Paclitaxel 60.0 mg/m2 / PM01183 5.0 mg FD (N=6) | Paclitaxel [80.0 mg/m2] / PM01183 [5.0 mg FD] (N=6) | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] (N=37) | Paclitaxel [80.0 mg/m2] / PM01183 [4.0 mg FD] / BEV 15 mg/kg (N=14)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (8) | 1 (1) | 2 (6) | 3 (13)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 5 (14) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (6)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (14)
Fatigue (General disorders) | 2 (11) | 3 (23) | 6 (42) | 6 (40) | 27 (153) | 10 (110)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (18) | 4 (22) | 1 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 4 (16) | 2 (19)
Pyrexia (General disorders) | 0 (0) | 2 (5) | 1 (1) | 2 (3) | 7 (17) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (19) | 1 (1)
Depression (Psychiatric disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (20)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (34) | 2 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (5) | 1 (2) | 6 (13) | 1 (3)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 4 (20) | 2 (8) | 11 (40) | 3 (13)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 2 (12) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 3 (5) | 2 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (4) | 8 (45) | 3 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 3 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 2 (11)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 3 (9) | 1 (1) | 7 (16) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (9) | 4 (17) | 5 (30) | 10 (22) | 3 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (19) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (26) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 2 (12) | 1 (3) | 0 (0) | 1 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (22) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (10) | 12 (59) | 2 (16)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (23)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (28) | 1 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0) | 3 (13) | 2 (6) | 1 (3)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (9) | 11 (33) | 6 (19)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (6) | 2 (6) | 13 (29) | 5 (13)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 4 (13) | 2 (16)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (7) | 1 (8)
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (5) | 2 (9) | 4 (16) | 24 (57) | 6 (29)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (10) | 0 (0) | 1 (1) | 1 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (5) | 3 (14) | 19 (29) | 3 (3)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (2) | 1 (6) | 5 (36) | 9 (47) | 5 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (11)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (7) | 2 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (3) | 2 (38)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 3 (17)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 2 (14) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (6) | 2 (6) | 10 (38) | 4 (20)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (18) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (23) | 2 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (5) | 0 (0)
Infusion site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Infusion site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Agitation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatitis acneiform (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less